CLINICAL TRIAL: NCT07167030
Title: Evaluation of the Effects of Digital Storytelling Applied to Primiparous Pregnant Women With Virtual Reality Glasses on Prenatal Attachment, Fear of Childbirth, Perception of Childbirth Self-Efficacy, and Non-Stress Test Results
Brief Title: Virtual Reality-Enabled Digital Storytelling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, RUKİYE DİKMEN, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1231
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Primiparous Pregnant Women
Keywords: Prenatal attachment; Fear of Childbirth; Birth Self-Efficacy; Virtual Reality; Digital Storytelling

STUDY DESIGN:
Intervention Model Description: Arm 1 Intervention Arm: Participants in the intervention group will receive digital storytelling modules using virtual reality (VR) headsets once a week for four weeks, starting at 28 weeks of gestation. Each module will include three topics (2-10 minutes). After each topic, there will be a rest period followed by an interactive session. The final two modules will be administered during the NST recording, and mother and baby status will be monitored. Each module, including the interactive session, will last 45-50 minutes. Participants will receive an educational brochure after the module and will be reminded via WhatsApp.
  Arm 2 Control Arm: Participants in the control group will receive routine care.
  Posttests (at the end of 36 weeks of gestation):
  * Prenatal Attachment Inventory
  * Wijma Birth Expectations/Experiences Questionnaire Version A
  * Short Version of the Labor Self-Efficacy Scale
  * Satisfaction Level Information Form for the VR Headset Application
  * NST Follow-up Form
  * Video
Who Masked: Participant
Masking Description: There is no other hidden side to this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Arm (Experimental): Participants in the intervention group will receive digital storytelling modules using virtual reality (VR) headsets once a week for four weeks, starting at 28 weeks of gestation. Each module will include three topics (2-10 minutes). After each topic, there will be a rest period followed by an interactive session. The final two modules will be administered during the NST recording, and mother and baby status will be monitored. Each module, including the interactive session, will last 45-50 minutes. Participants will receive an educational brochure after the module and will be reminded via WhatsApp.
  Posttests (at the end of 36 weeks of gestation):
  * Prenatal Attachment Inventory
  * Wijma Birth Expectations/Experiences Questionnaire Version A
  * Short Version of the Labor Self-Efficacy Scale
  * Satisfaction Level Information Form for the VR Headset Application
  * NST Follow-up Form
  * Video Immersion Scale
  Interventions: Behavioral: Virtual Reality Digital Storytelling
- Control Arm (No Intervention): Participants in the control group will receive routine care.
  Posttests (at the end of 36 weeks of gestation):
  * Prenatal Attachment Inventory
  * Wijma Birth Expectations/Experiences Questionnaire Version A
  * Short Version of the Labor Self-Efficacy Scale
  * NST Follow-up Form

INTERVENTIONS:
Behavioral: Virtual Reality Digital Storytelling — Participants in the intervention group will receive digital storytelling modules using virtual reality (VR) headsets once a week for four weeks, starting at 28 weeks of gestation. Each module will include three topics (2-10 minutes). After each topic, there will be a rest period followed by an interactive session. The final two modules will be administered during the NST recording, and mother and baby status will be monitored. Each module, including the interactive session, will last 45-50 minutes. Participants will receive an educational brochure after the module and will be reminded via WhatsApp.
  Arms: İntervention Arm

SUMMARY:
Current scientific literature on VR details primarily focuses on fear and anxiety during childbirth. Variables such as attachment, fear, and self-efficacy are often considered independently. Therefore, in addition to interventions focused on the prenatal period, a need arose for holistic audiovisual and technologically supported intervention models that simultaneously address multidimensional aspects of life, such as prenatal attachment, fear of childbirth, and perception of childbirth self-efficacy.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted to evaluate the effects of digital storytelling applied to primiparous pregnant women via virtual reality glasses on prenatal attachment, fear of childbirth, perception of childbirth self-efficacy, and non-stress test results. The study will consist of two groups: an experimental and a control group. Participants in the experimental group will access a digital storytelling training program via virtual reality glasses and receive information and guidance on topics such as prenatal attachment, fear of childbirth, and perception of childbirth self-efficacy. Participants in the control group will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women in their 28th week of pregnancy
* Between the ages of 18 and 40
* Experiencing a singleton pregnancy
* Applied to the Yozgat City Hospital Gynecology and Obstetrics Clinic and agreed to participate in the study
* Have a primary school education and can understand Turkish
* Have no serious vision or balance problems that would prevent the use of VR glasses
* Have not experienced any risky pregnancy problems (premature membrane rupture, preeclampsia, gestational diabetes, etc.)
* Have no identified fetal anomalies
* Have no psychiatric diagnosis

Exclusion Criteria:

* Pregnant women who cannot obtain a work permit and who do not agree to participate in the study will not be included in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals who are biologically female and experiencing their first reproduction are eligible to participate.
Enrollment: 112 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Prenatal Attachment Inventory | Time Frame: Pre-test (before intervention) Time Frame: Post-test (after intervention: 36th week of pregnancy, after the fourth module)
  The Prenatal Attachment Inventory (PAI) developed by Muller (1993) is used to assess the thoughts, feelings, and states experienced by women during pregnancy and to determine their attachment to their babies during the prenatal period (Muller, 1993). The Turkish validity and reliability study of the inventory, conducted by Yılmaz and Beji (2013), consists of 21 items. Each item is a four-point Likert-type scale, ranging from 1 to 4. A minimum score of 21 and a maximum score of 84 can be obtained from the scale. Increasing scores indicate increased attachment. The scale's validity and reliability performance was found to be 0.84, with a Cronbach's alpha of 0.10.
Wijma Childbirth Expectation/Experience Questionnaire Version A (W-DEQ-A) | Time Frame: Pre-test (before intervention) Time Frame: Post-test (after intervention: 36th week of pregnancy, after the fourth module)
  Developed by Wijma et al. (1998) to assess the level of fear of childbirth experienced by pregnant women, the scale was adapted into Turkish by Körükcü (2009). Version A of the W-DEQ is a 33-item scale. Responses are numbered from 0 to 5 and are on a six-point Likert-type scale. The minimum score is 0, and the maximum score is 165. A high total score indicates a high level of fear. In the validity and reliability study of the scale, Cronbach's Alpha was found to be 0.89 (Körükcü, 2009).
Short Version of the Labor Self-Efficacy Scale | Time Frame: Pre-test (before intervention) Time Frame: Post-test (after intervention: 36th week of pregnancy, after the fourth module)
  The Turkish adaptation of the scale, developed to measure women's self-efficacy for childbirth, was conducted by Ersoy (2011). The scale consists of two sub-dimensions: competence and outcome expectation, and a total of 32 questions. Scores for each sub-dimension range from 16 to 160. As the score on each sub-dimension increases, the competence and outcome expectation for childbirth increases. The Likert-type scale is scored from 1 to 10. In the outcome expectation sub-dimension of the scale, 1 represents "not at all useful," and 10 represents "very useful." In the competence expectation sub-dimension, questions 1 to 13 are scored as 1 "completely confident," 10 represents "not at all confident," and the remaining questions are scored as 1 "not at all confident," and 10 represents "completely confident." The first 13 questions in the competence expectation sub-dimension of the scale are reverse-scored. The total score obtained from the scale ranges from 32 to 320. As the score on the

SECONDARY OUTCOMES:
NST Follow-up Form | Time Frame: 34th weeks of pregnancy (during the last two modules) Time Frame: 36th weeks of pregnancy (during the last two modules)
  This form consists of sections containing the emotional state and NST findings experienced by pregnant women during the NST procedure. The NST results in the NST Follow-up Form will be evaluated and recorded by the researcher.

OTHER OUTCOMES:
Video Immersion Scale (VIS) | Time Frame: Post-intervention (post-intervention: 36th week of pregnancy, after the fourth module)
  The Video Immersion Scale, developed by Visser et al. (2016), was adapted into Turkish by Deryakulu et al. (2019). The scale consists of five factors and a total of 15 items. The Cronbach's alpha internal consistency coefficients calculated for the subfactors and the entirety of the Video Immersion Scale, which is a seven-point Likert-type scale, are as follows: Factor 1 (Attention) 0.57; Factor 2 (Narrative World Immersion) 0.73; Factor 3 (Identity) 0.87; Factor 4 (Empathy) 0.78; Factor 5 (Emotion) 0.69; and for the entire scale, 0.90. In this study, the Cronbach's alpha reliability coefficients for the factors were, respectively, Factor 1 (Attention) 0.57; Factor 2 (Entering the narrative world) was calculated as 0.71; Factor 3 (Identity) as 0.70; Factor 4 (Empathy) as 0.72; Factor 5 (Emotion) as 0.78; and 0.81 for the entire scale.
Virtual Reality Glasses Application Satisfaction Level Information Form | Time Frame: Post-intervention (post-intervention: 36th week of pregnancy, after the fourth module)
  This form will include questions prepared by researchers to determine satisfaction with the video watched with virtual reality glasses.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant confidentiality and as data was collected only for this study.